CLINICAL TRIAL: NCT03265262
Title: Evaluation of Technical and Predictive Value of the Basophil Activation Test for Food Allergy Diagnosis in Children
Brief Title: The Basophil Activation Test as a Diagnostic Tool in Pediatric Food Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-26
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: FOOD ALLERGY
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children receiving OFC during a diagnost (Experimental): paediatric patients attending food allergy
  Interventions: Diagnostic Test: The basophil activation test (BAT)

INTERVENTIONS:
Diagnostic Test: The basophil activation test (BAT) — Single sample: 5 mL of venous blood

SUMMARY:
Background: The need for an oral food challenge (OFC) surrogate is growing in line with the continuous increase in the prevalence and severity of paediatric food allergy. The basophil activation test (BAT) has recently been reported as a promising tool for predicting the outcome of OFC in children.

Objective: We make the hypothesis that BAT might improve the sensitivity of food allergy diagnosis and spare part of current OFC in paediatric patients attending allergy departments in Marseille APHM University hospitals.

Methods: BAT will be performed in parallel with OFC in 100 paediatric patients receiving OFC during a diagnostic or follow-up procedure.

Expected results: Good concordance of BAT and OFC results leading to potential OFC replacement by BAT in at least 50% of the study population

ELIGIBILITY:
Inclusion Criteria:

* Age 0 - 18 years
* Attending La Timone Paediatric Hospital for OFC
* Social insurance
* Parents and if possible child have received information and signed the consent form

Exclusion Criteria:

* Patients not receiving an OFC
* Lack of social insurance
* Inability to understand the study information
* Unwilling to participate

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
BAT positive and negative predictive values as compared with OFC | 2 years
  BAT versus OFC

SECONDARY OUTCOMES:
BAT quantitative results as compared with the minimal reacting dose for OFC | 2 years
  BAT versus OFC

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Arif-Lusson R, Agabriel C, Carsin A, Cabon I, Senechal H, Poncet P, Vitte J, Busnel JM. Streamlining basophil activation testing to enable assay miniaturization and automation of sample preparation. J Immunol Methods. 2020 Jun-Jul;481-482:112793. doi: 10.1016/j.jim.2020.112793. Epub 2020 May 6. PMID 32387696